CLINICAL TRIAL: NCT05417464
Title: Evaluation and Validation of a Monitoring, Screening and Management Strategy for Conductive Disorders After TAVR (EVATAVI)
Brief Title: Evaluation and Validation of Management Strategy for Conductive Disorders After TAVR (EVATAVI)
Acronym: EVATAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0646
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Valvular Heart Disease
Keywords: Aortic Valve,; Aortic Valve Stenosis,; Heart Valve Prosthesis Implantation,; Transcatheter Aortic Valve Replacement,; Telemetry,; Intensive care
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: This is a non-comparative prospective interventional study, involving the human category, which aims to evaluate the efficacy and safety of a flowchart for screening, monitoring and management of conductive disorders after TAVR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Management of conductive disorders after TAVR (Other): Evaluation of efficacy and safety of a flowchart for screening, monitoring and management of conductive disorders after TAVR
  Interventions: Other: Use of flowchart

INTERVENTIONS:
Other: Use of flowchart — Use of flowchart for screening, monitoring and management of conductive disorders after TAVR

SUMMARY:
Considering decrease of major complications and improvement of procedural results, conductive disorders currently remain the main issue after TAVR (Transcatheter aortic valve replacement).

While pacemaker implantation rate was about 10-15%, new onset LBBB (Left bundle branch block) was observed in 30 % of patients after TAVR but resolved at discharge in the majority of them, with less than 20% progressed to complete AV (atrioventricular) block requiring permanent pacing at hospital discharge.

Higher implantation and improvement of the devices were associated with decline of pace maker implantation rate over the years in experienced teams.

While guidelines do not give definite recommendation regarding conductive disorder management and pacemaker indication, a strategy of selective telemetry monitoring (TM) after TAVR according to the risk of conductive disorders may be proposed to limit indication and lenght of stay of intensive care unit admission (ICU), allowing direct admission of lower risk patients in general cardiology ward (GCW) without TM, to decrease the duration of TM when a conductive disorder is stable or regressive and finally to decrease the rate of pacemakers implantation.

Potential benefit may also include limitation of ICU overload in high volume TAVR centers, investigators can also expect shorter hospitalization duration, with potential economic impact, in line with the development of algorithms for fast track procedures.

Therefore the main objective of our prospective study was to evaluate feasibility and safety of a strategy of management of conductive disorders after TAVR based on an algorithm of diagnosis, monitoring and therapeutic strategies based on ECG analysis.

DETAILED DESCRIPTION:
TAVR is now the reference method for the treatment of severe aortic stenosis in the elderly population. Regarding its good results, indications have recently been extended to younger, lower-risk patients. With the decrease in serious complications, severe conductive disorders requiring the implantation of a pacemaker have thus become the main complications of TAVR.

Despite the experience of operators and modified implantation techniques and in absence of specific recommendations, the rate of pacemaker implantation after a TAVR procedure levels off between 10% and 20% regardless of the prosthesis used and with highly variable rates depending on the center.

In the vast majoriy of cases, the conductive disorders only justify the monitoring of patients in ICU after the procedure,

However, majority of conductive disorders will be regressive or stable and will not justify a permanent pacemaker implantation. Furthemore, this systematic monitoring contributes to unnecessarily overcrowding of these medical structures.

Investigators thus put forward the hypothesis that by using a defined strategy for screening and monitoring conductive disorders occurring after a TAVR procedure, and by taking into account the recommendations on indication of definitive cardiac pacing, it would be possible to rationalize both the indications, the duration of monitoring (by telemetry/CICU or conventional sector) and the definitive pacemaker indication.

Investigators thus hope, thanks to this rationalized strategy, to reduce the indications and durations of monitoring by telemetry or CICU after a TAVR and to shorten the durations of overall hospitalization, but also to reduce the indication for permanent cardiac pacing without risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who benefits from femoral TAVR regardless of the type of valve.
* Age ≥ 18 years old.

Exclusion Criteria:

* Patients who require CICU monitoring for a reason other than conduction disorders
* Patients with pacemaker or defibrillator
* Pregnant or breastfeeding women
* Patient refusing or unable to give consent: patient under guardianship or curator, mentally retarded, dementia, language barrier
* Patient not affiliated with an SS scheme
* Patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-02-21 (Estimated); Study Completion 2024-03-21 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a serious conductive disorder | Between inclusion and 1 month after TAVR procedure
  Occurrence of a serious conductive disorder (one among the following : syncope, malaise, sudden death, heart failure) outside the CICU (whether the patient was there admitted initially or not)
Occurrence of a serious conductive disorder requiring specific management | Between inclusion and 1 month after TAVR procedure
  Occurrence of a serious conductive disorder requiring specific management (one among the following : drug treatment, need for a transient or permanent pacemaker), outside the CICU (whether the patient was there admitted initially or not)

SECONDARY OUTCOMES:
Incidence and type of conductive disorders requiring transfer to CICU (cardiac intensive care unit) | Between inclusion and 1 month after TAVR procedure
Pourcentage of Pacemaker implantation | Between inclusion and 1 month after TAVR procedure
Time of onset of conductive disorders requiring a pacemaker (immediate, hospital phase, after discharge from hospital) | Between inclusion and 1 month after TAVR procedure
Description of the evolution of conductive disorders that have not been the subject of pacemaker insertion (hospitalization) | Between inclusion and 1 month after TAVR procedure
  Number of conductive disorders that lead to patient's rehospitalization
Description of the evolution of conductive disorders that have not been the subject of pacemaker insertion (death) | Between inclusion and 1 month after TAVR procedure
  Number of conductive disorders that lead to patient's death
Death | Between inclusion and 1 month after TAVR procedure
Clinical status at one month (NYHA (New York Heart Association) | Between inclusion and 1 month after TAVR procedure
Death within the first month after TAVR | Between inclusion and 1 month after TAVR procedure
Duration of hospitalization in CICU | Between inclusion and 1 month after TAVR procedure
Duration of hospitalization in sector | Between inclusion and 1 month after TAVR procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided